CLINICAL TRIAL: NCT00062699
Title: A Phase IV, Prospective, Randomized, Active-Controlled, Double-Blind, Double-Dummy, Multi-Center Study to Evaluate the Survival Benefits of Zemplar Relative to Calcijex in Subjects With Stage V Chronic Kidney Disease on Hemodialysis
Brief Title: Evaluate the Survival Benefits of Zemplar Versus Calcijex in Subjects w/ Stage V Chronic Kidney Disease on Hemodialysis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-516
Record Dates: First submitted 2003-06-11; First posted 2003-06-13 (Estimated); Last update posted 2006-08-02 (Estimated); Status verified 2006-07

CONDITIONS: End-Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — paricalcitol; Calcitriol

INTERVENTIONS:
Drug: Zemplar (paricalcitol injection)
Drug: Calcijex

SUMMARY:
To evaluate the survival benefit associated with Zemplar therapy as compared to Calcijex for the treatment of secondary hyperparathyroidism in subjects with Stage V chronic kidney disease on hemodialysis as measured by time to death.

ELIGIBILITY:
Stage V Chronic Kidney Disease Patients on Hemodialysis requiring treatment for secondary hyperparathyroidism with vitamin D therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200
Dates: Start 2003-04

PRIMARY OUTCOMES:
Time to Death

SECONDARY OUTCOMES:
Time to Death attributable to cardiovascular disease
Number of hospitalizations for any cause
Number of hospitalizations due to cardiovascular disease
Number of days hospitalized for any cause
Number of days hospitalized due to cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 1-800-633-9110, Study Director — Abbott
Locations (59):
- United States (59):
  - Tuscaloosa Nephrology Associates, Tuscaloosa, Alabama
  - Gambro Healthcare - Inglewood, Inglewood, California
  - Gambro Healthcare - Los Angeles, Los Angeles, California
  - Apex Research of Riverside, Riverside, California
  - East Bay Nephrology Medical Group, San Pablo, California
  - Nephrology Educational Services and Research, Inc., Tarzana, California
  - Lowry DaVita Dialysis Unit, Denver, Colorado
  - Stamford Nephrology, Stamford, Connecticut
  - Capital Dialysis Unit, Washington D.C., District of Columbia
  - Capitol Dialysis, Washington D.C., District of Columbia
  - Dupont III, P.C., Washington D.C., District of Columbia
  - Capital Dialysis Northwest, Washington D.C., District of Columbia
  - Renal Associates of Boca Raton, Boca Raton, Florida
  - Associates in Nephrology, Fort Myers, Florida
  - Orlando Nephrology, Winter Garden, Florida
  - Nephrology Associates, P.C., Augusta, Georgia
  - Nephrology Center of America - Augusta, Augusta, Georgia
  - Nephrology Center of America - South Augusta, Augusta, Georgia
  - Nephrology Center of America - Grovetown, Grovetown, Georgia
  - Nephrology Center of America - Vidalia, Vidalia, Georgia
  - Northwestern University - Division of Nephrology, Chicago, Illinois
  - Renal Care Group, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Louisiana State University Health and Sciences Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Uptown Dialysis Center, New Orleans, Louisiana
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Paul Light, University of Maryland, Baltimore, Maryland
  - Gambro Healthcare - Whitesquare Dialysis Center, Baltimore, Maryland
  - Gambo Healthcare - JB Zachary Dialysis Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Gambro Healthcare - Dundalk Dialysis Center, Dundalk, Maryland
  - Kidney Center of Frederick, Frederick, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Nephrology Foundation of Brooklyn, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Gates Circle Dialysis, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Chinatown Dialysis Center, New York, New York
  - Lower Manhatten Dialysis Center, New York, New York
  - Columbia University Dialysis Center, New York, New York
  - Orchard Park Dialysis, Orchard Park, New York
  - Suburban Dialysis Center, Williamsville, New York
  - The Rogosin Institute, Woodside, New York
  - Dialysis Clinic Inc, Cincinnati, Ohio
  - Northwest Renal Clinic, Inc., Portland, Oregon
  - Doylestown Dialysis Center, Doylestown, Pennsylvania
  - Renal Care of Erie, Erie, Pennsylvania
  - Arlington Nephrology, PA, Arlington, Texas
  - UT Southwestern Medical School at Dallas, Nephrology Research Outpatient Clinic, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Jefferson Nephrology, Charlottesville, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Gambro Healthcare, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia